CLINICAL TRIAL: NCT01889849
Title: Comparative Pharmacokinetics and Pharmacodynamics, and Safety of Two Products Containing Recombinant Human Interferon Alpha-2 Conjugated to Polyethylene Glycol in Healthy Volunteers - Phase 1.
Brief Title: Comparative Pharmacokinetics and Pharmacodynamics of Peginterferon BIP48 and 40kDa in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASCLIN 003/2009
Record Dates: First submitted 2013-06-19; First posted 2013-07-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Viral Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BIP48 (Experimental): Will be recruited for the study 32 volunteers, all of whom will receive two products in two stages separated by at least 4 weeks. Volunteers will be randomized into 2 groups of 16 and at the time of the intervention, the volunteer will receive product application labeled with its corresponding number. The second step in the product administered will necessarily be one that contains the number and it was not administered in the first step.
  Interventions: Drug: BIP 48; Drug: Pegasys
- Pegasys (Active Comparator): Will be recruited for the study 32 volunteers, all of whom will receive two products in two stages separated by at least 4 weeks. Volunteers will be randomized into 2 groups of 16 and at the time of the intervention, the volunteer will receive product application labeled with its corresponding number. The second step in the product administered will necessarily be one that contains the number and it was not administered in the first step.
  Interventions: Drug: BIP 48; Drug: Pegasys

INTERVENTIONS:
Drug: BIP 48 — Volunteers will be randomized into two groups, and each one will receive the two products in two stages separated by at least 4 weeks.
  Other Names: Peginterferon alfa 2b 48kDA
Drug: Pegasys — Volunteers will be randomized into two groups, and each one will receive the two products in two stages separated by at least 4 weeks.
  Other Names: Peginterferon alfa 2a 40kDA

SUMMARY:
This research protocol "Comparative pharmacokinetics and pharmacodynamics of peginterferon Bacterial Intravenous Protein 48 kilodaltons (BIP48) and 40 kilodaltons (40kDa) in healthy volunteers." This is a Phase I clinical trial which will compare pharmacokinetic and pharmacodynamic parameters, and safety of two products: peginterferon alfa-2a (PEGASYS ®) and BIP48. It will be a double-blind, randomized crossover with a rest period (wash-out) of 4 weeks. The study population will be 32 healthy male volunteers to whom will be administered a single dose of 180 microgram of each product, subcutaneously. The study will have a total duration of 14 days in each treatment step. The serum concentration of PEG-interferon for both products, measured by enzyme immunoassay (EIA) and by antiviral activity of PEG-interferon, is the main variable.For this purpose 15 samples of each volunteers will be needed. Clinical and laboratory variables, useful as pharmacodynamics parameters Beta-2 microglobulin (β2M) - 2'5'oligoadenylate synthetase - oligoadenylate synthetase (OAS)- and neopterin) and safety evaluation, will be measured.

DETAILED DESCRIPTION:
Double-blind study, ie, the volunteers and the study team will not be aware of the product administered. As the presentations of the two products are different, only the professional who will administer the injections will not be blinded, and will not have contact with volunteers or members of the study team after applying the medication.

ELIGIBILITY:
Inclusion Criteria:

* No history of chronic diseases;
* Preserved oral health;
* No history of acute illness in the last 30 days;
* Absence of significant clinical symptoms and signs on physical examination;
* laboratory tests within normal limits;
* imaging tests within normal limits;
* Seronegative tests for HIV and B and C Hepatitis; Signing the consent form;
* Male;
* Age between 18 and 35 years;
* Body mass index between 19 and 26 (weight in kg / height in meters squared).

Exclusion Criteria:

* Patients with hypersensitivity to Interferon alpha, Escherichia coli-derived products, polyethylene glycol (macrogol), or any constituent salts of these preparations.
* Individuals treated with some type of interferon at any time, prior to the present research.
* History of chronic diseases such as autoimmune diseases, liver failure, decompensated cirrhosis, heart disease, renal failure, diabetes mellitus, thyroid diseases, hemoglobinopathies, cytopenias, history of psychiatric disease, retinopathy, optic neuritis.
* History of acute viral disease in the last 30 days;
* Current use of medications that alter immunity: corticosteroids, immunosuppressants;
* History of known allergy to drugs, including interferon or to any component of the product (at the discretion of the investigator);
* Having undergone surgery during the 6 months prior to study entry; Had donated blood three months prior to study entry;
* History of alcoholism or current use of alcohol;
* Use of other illicit drugs in the past 6 months;
* Participation in a clinical study with previous therapeutic intervention in the year prior to inclusion.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety Assessment | 14 days + least 4 weeks (rest period between each administration) + 14 days
  Evaluation of safety will be estimated by the analysis of clinical chemistry and hematology (CBC and transaminase) prior to study initiation and at 24, 48, 72, 96, 120, 168 and 336 hours after administration of peginterferon alpha, in each treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Dornelles Picon, Doctorate, Principal Investigator — Immunobiological Technology Institute (Bio-Manguinhos)
Locations (1):
- Bio-Manguinhos/Fiocruz, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] da Silva AMV, Alvarado-Arnez LE, Azamor T, Batista-Silva LR, Leal-Calvo T, Bezerra OCL, Ribeiro-Alves M, Kehdy FSG, Neves PCDC, Bayma C, da Silva J, de Souza AF, Muller M, de Andrade EF, Andrade ACM, Dos Santos EM, Xavier JR, Maia MLS, Meireles RP, Cuni HN, Sander GB, Picon PD, Matos DCS, Moraes MO. Interferon-lambda 3 and 4 Polymorphisms Increase Sustained Virological Responses and Regulate Innate Immunity in Antiviral Therapy With Pegylated Interferon-Alpha. Front Cell Infect Microbiol. 2021 Jul 7;11:656393. doi: 10.3389/fcimb.2021.656393. eCollection 2021. PMID 34307188
- [Derived] Costa MB, Picon PD, Sander GB, Cuni HN, Silva CV, Meireles RP, Goes ACMA, Batoreu NM, Maia MLS, Albuquerque EM, Matos DCS, Saura PL. Pharmacokinetics comparison of two pegylated interferon alfa formulations in healthy volunteers. BMC Pharmacol Toxicol. 2018 Jan 4;19(1):1. doi: 10.1186/s40360-017-0192-z. PMID 29301580